CLINICAL TRIAL: NCT02076035
Title: A Prospective Study to Analyze, in a Population Undergoing to a Periduroscopy Approach, the Correlation Between Outcome of Procedure and Histological-biochemical Neuroinflammation and Genetic Factors
Brief Title: Periduroscopy: Correlation Between the Outcome of Procedure and Histological-biochemical, Neuroinflammation and Genetic Factors.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Parma (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Guido Fanelli, Professor, University of Parma
Other Study IDs: Pain-Omics Periduroscopy
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; periduroscopy; genetic; genomic; inflammation
MeSH Terms: conditions — Low Back Pain; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3 whole blood samples will be collected: before epiduroscopy, immediately after it and after a month for genetic analyses and cytokine dosage. An epidural bioptic sample will be performed according to usual clinical practice
Oversight: Data Monitoring Committee: No

SUMMARY:
It is still unknown the pathogenesis of low back pain and a lot of hypothesis were discussed for a long time. Because non-invasive imaging modalities greatly underestimate the prevalence of epidural pathogenesis an endoscopic examination of the epidural space has been advocated as both a diagnostic and therapeutic modality. It seems that immune-inflammatory factors play a more substantial role in pain status. Myeloscopic investigation have shown how morphological pictures of the epidural area in patients with chronic low back pain (CLBP) are much more complex and heterogeneous than what can be identified with traditional investigation suggesting a biochemical involvement. Endoscopy of the epidural space (epiduroscopy) is a minimally invasive technique, used to directly visualize pathological features inside of the lumbar spinal canal to locate tissues responsible of eliciting pain and the presence of any pathological structures within the vertebral channel, such as fibrous adherences, inflammatory processes, severe fibrosis and/or stenoses, in order to realize an effective therapeutic approach in a lot of different CLBP status as those due to spinal stenoses or failed back surgery syndrome. To deepen the molecular causes of interindividual variability of epiduroscopy outcomes in terms of decrease of pain, it is useful to analyze the DNA variants encoding IL6 and IL1 cytokines and to relate them with gene expression levels and with the cytokine dosage. By this technique, it is possible to analyze in the biopsy of the epidural tissue the specific expression of the cytokines: there is already evidence that inflammatory factors may be involved in the genesis of LBP. At this regards, it would be really important to compare systemic cytokine levels before the epiduroscopy with those detected immediately post procedure and after one month, to understand if the cytokines could play a key role and be a biomarker of the epiduroscopy outcome.

Concerning DNA polymorphisms, it has been demonstrated, in many disease-state meta-analyses, that the IL6 variant rs1800795 affect gene transcription and influences the IL-6 levels. Moreover, interleukin 1 (IL-1) is a major factor controlling the inflammatory response. The IL-1 gene family includes the IL-1α, IL-1β and the IL-1 receptor antagonist (IL-1Ra) genes that mediate immune and inflammatory responses. SNPs in IL-1α, IL-1β and IL1Ra modify bone mineral density promoting intervertebral disc disease (IDD). The simultaneous carriage of the IL-1bT3954 and the IL-1Ra A1812 alleles significantly enhances the risk of low back pain (LBP) occurrence, the number of days with pain, and the number of days with limitations in daily activities due to pain.

A recent study suggested that methylation status of a single CpG site in the IL6 promoter is related to IL6 messenger RNA levels and that lower methylation contributes to the risk of developing Rheumatoid Arthritis.

The investigators will try to identify if it there is a correlation with success of the epiduroscopy approach in terms of freedom from pain with genic expression and cytokine dosage.

Finally, the investifators will compare the cytokine gene expression and the DNA methylation status of IL6 promoter in patients with favorable outcome and in no responders, to study the role in gene expression.

This study is addressed to detect if the genetic variability might be used in near future in clinical setting, to predict the success of epiduroscopy.

DETAILED DESCRIPTION:
It is still unknown the pathogenesis of low back pain and a lot of hypothesis were discussed for a long time. Because non-invasive imaging modalities greatly underestimate the prevalence of epidural pathogenesis an endoscopic examination of the epidural space has been advocated as both a diagnostic and therapeutic modality.

It seems that immune-inflammatory factors play a more substantial role in pain status. Myeloscopic investigation have shown how morphological pictures of the epidural area in patients with chronic low back pain (CLBP) are much more complex and heterogeneous than what can be identified with traditional investigation suggesting a biochemical involvement.

Endoscopy of the epidural space (epiduroscopy) is a minimally invasive technique, which can be used to directly visualize pathological features inside of the lumbar spinal canal to locate tissues responsible of eliciting pain and realize an effective therapeutic approach in a lot of different CLBP status as those due to spinal stenoses or failed back surgery syndrome.

Minimally invasive endoscopic exploration of the lumbar epidural cavity in patients suffering from chronic low back pain has been used to identify the presence of any pathological structures within the vertebral channel, such as fibrous adherences, inflammatory processes, severe fibrosis and/or stenosis. The need to visually inspect the epidural space originally arose as conventional imaging, such as magnetic resonance imaging (MRI), has been shown to be significantly less sensitive in identifying epidural pathology compared with direct visualization. In a cohort of failed back surgery syndrome (FBSS) patients, 80% of those having severe epidural fibrosis diagnosed with epiduroscopy had a normal MRI examination. More, when used to identify the exact spinal level of painful pathology, neither clinical examination nor MRI evaluation strongly correlated with the endoscopy findings.

The combination of a disposable and easily steerable small video-guide, high-resolution optics and specifically designed tools such as mechanical dissectors, electric knife and graspers, makes this technique as a valid option to diagnose and treat epidural pathology in the lumbar region.

To deepen the molecular causes of interindividual variability of epiduroscopy outcomes in terms of decrease of pain, it is useful to analyze the DNA variants encoding IL6 and IL1 cytokines and to relate them with gene expression levels and with the cytokine dosage. By this technique, it is possible to collect a biopsy of the epidural tissue (usually performed during epiduroscopy) analyzing the specific expression of the cytokines: there is already evidence that inflammatory factors may be involved in the genesis of LBP. At this regards, it would be really important to compare systemic cytokine levels before the epiduroscopy with those detected immediately post procedure and after one month, to understand if the cytokines could play a key role and be a biomarker of the epiduroscopy outcome.

Concerning DNA polymorphisms, it has been demonstrated, in many disease-state meta-analyses that the IL6 variant rs1800795 affect IL6 gene transcription and influences the IL-6 levels ensuring the statistical robustness of the associations.

Moreover, interleukin 1 (IL-1) is a major factor controlling the inflammatory response. The IL-1 gene family includes the IL-1α, IL-1β and the IL-1 receptor antagonist (IL-1Ra) genes that mediate immune and inflammatory responses. The IL-1Ra molecule has been shown to be a powerful anti-inflammatory agent inhibiting the activities of IL-1 α and IL-1β. Moreover, SNPs in IL-1α, IL-1β and IL1Ra modify bone mineral density promoting intervertebral disc disease (IDD). Literature data showed that the simultaneous carriage of the IL-1bT3954 and the IL-1Ra A1812 alleles significantly enhances the risk of low back pain (LBP) occurrence, the number of days with pain, and the number of days with limitations in daily activities due to pain.

The investigators will try to identify if it there is a correlation with success of the epiduroscopy approach in terms of freedom from pain with genetic and cytokine expression patterns.

Finally, the investigators will compare the cytokine gene expression and the DNA methylation status of IL6 promoter in patients with favorable outcome and in no responders, to study its role in gene expression. In fact, a recent study suggested for the first time that methylation status of a single CpG site in the IL6 promoter is related to IL6 messenger RNA levels and that lower methylation contributes to the risk of developing Rheumatoid Arthritis.

This study is addressed to detect if the genetic variability might be used in near future in clinical setting, to predict the success of epiduroscopy.

The main aim of this study consists in identifying whether a particular genotype associated with inflammation is able to detect which patients will have a positive epiduroscopy outcome, in terms of decrease of pain.

To achieve it, the investigators will investigate the frequency of some IL1 and IL6 gene polymorphisms: we will analyze and compare IL1β, IL1Ra, IL6 and IFNγ blood cells gene expression (before, immediately post the epiduroscopy and after one month) with that obtained by epiduroscopy biopsy cells.

The investigators will also measure IL1β, IL1Ra, IL6 and IFNγ levels from patient serum before the epiduroscopy, immediately post the procedure and after 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 75 years
* Patients undergone periduroscopy procedure according to good clinical practice.
* Written informed consent signed

Exclusion Criteria:

* Subjects with evidence of clinically unstable disease (without stable treatment that needs continuous pharmacological and drugs dosage changes; physicians requiring further assessments; at instance not-responder hypertension to the pharmacological treatment with pressure values constantly alterated despite the therapy)
* Subjects with a severe psychiatric disorder diagnosed by a psychiatrist and / or neurologist, that are/have been under a pharmacological treatment and under specialist control with particular contraindications to invasive treatments
* Mental impaired patients
* History of spinal fracture
* Spinal tumor or infection of column;
* Visual alterations (glaucoma, diabetic retinopathy)
* Brain vascular disease
* Primary or secondary chronic headache
* For women: positive pregnancy test or pregnancy.
* Coagulopathy (INR>1.5)
* Refusal to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll a well phenotyped cohort of patients with chronic low back pain, sub-grouped into categories: spinal stenosis (congenital or acquired) and failed back surgery syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
genetic outcome | 36 months
  the frequency of rs1800795 in the promoter of the IL6 gene

SECONDARY OUTCOMES:
genomic outcome | 36 months
  other known variants related to inflammation in IL1β and IL6 loci
inflammation outcome | 36 months
  IL-6, IL-1β, IL1Ra and INFγ serum concentration before, immediately post epiduroscopy and after 1 month
gene expression outcome | 36 months
  IL-6, IL-1β, IL1Ra and INFγ gene expression in blood cells obtained before, immediately post epiduroscopy and after 1 month
biopsy tissue outcome | 36 months
  IL-6, IL-1β, IL1Ra and INFγ gene expression in biopsy tissue cells
methylation outcome | 36 months
  the methylation of the promoter of IL6

CONTACTS AND LOCATIONS:
Locations (1):
- University of Parma, Parma, Parma, Italy